CLINICAL TRIAL: NCT06871423
Title: Magic Bowl VR Analgesia
Brief Title: The Effect of Virtual Reality on Pain and Memory.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Hunter Hoffman, Director, Virtual Reality Research Center at the Human Photonics Lab; Research Scientist:Dept of Mechanical Engineering, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VRAnalgesia2022
Record Dates: First submitted 2025-03-01; First posted 2025-03-12 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy Adult
Keywords: virtual reality; pain; distraction
MeSH Terms: conditions — Pain | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Intervention Model Description: Using a repeated measures within-subject crossover design with treatment order randomized, with healthy volunteers,
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Virtual Reality (No Intervention): No Virtual Reality during painful stimuli
- Immersive VR (Experimental): immersive virtual reality during painful stimuli
  Interventions: Behavioral: distraction

INTERVENTIONS:
Behavioral: distraction — distraction via virtual reality game named "Waltz of the Wizards" aka magic bowl.
  Arms: Immersive VR

SUMMARY:
The effect of Virtual Reality on pain and memory.

DETAILED DESCRIPTION:
The primary outcome measure was the participants' accuracy of remembering the pattern of a total of five pain stimuli per set. Using the Quantitative Sensory Testing "method of limits", each participant selected a temperature they found "painful but tolerable" that they were willing to receive several more times, later in the study. They then received a sequence of five brief stimuli to their wrist, with a brief inter-stimulus interval between each stimulus.

ELIGIBILITY:
Inclusion Criteria:

* must be English speaking (but English does not necessarily need to be native/first language).
* must be willing to follow our UW approved instructions,

Exclusion Criteria:

* Not capable of indicating pain intensity
* Not capable of filling out study measures
* Non-English-speaking
* Extreme susceptibility to motion sickness
* Seizure history
* Unusual sensitivity or lack of sensitivity to pain
* Sensitive skin
* sensitive feet
* migraines
* cold symptoms
* Diabetes
* Or if you are under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Pain Memory Recall Test | After each brief pain stimulus set, participants performed a brief distractor task before completing the Pain Memory Recall Test. The Pain Memory Recall Test was completed within 5 minutes after each brief thermal stimulus set.
  After each brief thermal stimulus set, participants were asked to recall the exact pattern of the most recent sequence of 5 brief thermal stimuli, recalled in exact order, via our five question "pain memory recall test" (min = 0%, max -= 100% correct). Lower % correct scores mean less accurate memory (poorer outcome).
Participants subjective rating of the accuracy of their memory for painful stimuli | measured within 10 minutes after each pain stimulus set
  Using a graphic rating scale, on a scale from zero (min) to 10 (max), participants rated how accurately they could remember their pain during No Virtual Reality vs during Virtual Reality. Higher scores indicated higher accuracy and more positive outcome.

SECONDARY OUTCOMES:
Presence ratings using Graphic Rating Scales | measured within 10 minutes after participant was in virtual reality
  Participants rated their illusion of "being there" in the computer generated world, as if it was a place they were visiting, on a scale from zero to 10, where zero = none at all and 10 = "completely there".

CONTACTS AND LOCATIONS:
Overall Officials: Hunter G Hoffman, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All data is already de-identified. Only de-identified data will be shared. The datasets used and/or analyzed during the current study will be made available from the corresponding author on reasonable request. All de-identified IPD that underlie our results in a publication will be shared.
Time Frame: Beginning 3 months after the publication of the results, and ending 3 years after the publication of results
Access Criteria: All data is already de-identified. Only de-identified data will be shared. The datasets used and/or analyzed during the current study will be made available from the corresponding author on reasonable request. All de-identified IPD that underlie our results in a publication will be shared.